CLINICAL TRIAL: NCT03697564
Title: Open Label Randomized Phase II Trial of Nivolumab + Cabiralizumab (BMS-986227, FPA008) + Gemcitabine in Patients With Stage IV Pancreatic Cancer Achieving Disease Control in Response to First-line Chemotherapy (GemCaN Trial)
Brief Title: Nivolumab + Cabiralizumab + Gemcitabine in Patients With Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hitendra Patel (Other)
Collaborators: Stand Up To Cancer (Other); Lustgarten Foundation (Other)
Responsible Party: Sponsor-Investigator, Hitendra Patel, Associate Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181395
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Stage IV
Keywords: Pancreating Cancer; Cancer; Stage IV; gemcitabine; nivolumab; cabiralizumab; BMS-986227; FPA008; GemCaN; Stand Up to Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Nivolumab; cabiralizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- gemcitabine +nivolumab + cabiralizumab (Experimental): gemcitabine +nivolumab + cabiralizumab
  Interventions: Drug: Gemcitabine; Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO]; Drug: Cabiralizumab

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 IV on days 1, 8, and 15 Q4W
  Other Names: Gemzar and Infugem
Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO] — 480mg IV on Day 1 Q4W
  Other Names: Opdivo
Drug: Cabiralizumab — 4mg/kg IV on day 1 and 15 Q4W
  Other Names: FPA 008

SUMMARY:
The purpose of this study is to see if the combination of nivolumab + cabiralizumab + gemcitabine can give prolonged disease control in patients with advanced pancreatic cancer compared to gemcitabine alone.

DETAILED DESCRIPTION:
The purpose of this study is to see if the combination of nivolumab + cabiralizumab + gemcitabine can give prolonged disease control in patients with advanced pancreatic cancer compared to gemcitabine alone.

Cabiralizumab is an antibody (a type of protein) that binds to a molecule called CSF-1r. CSF-1r is a molecule present on different types of cells in your immune system that controls parts of your immune system. Blocking CSF-lr could potentially stop the cancer cells which it appears on from escaping the immune system, which could then act to kill the cancer cells.

Nivolumab is an anti-PD-1 antibody that boost the body's immune system. It works by attaching to and blocking a molecule on white blood cells called PD-1. PD-1 is a protein that is present on different types of cells in your immune system and controls parts of your immune system by shutting it down. Antibodies that block PD-1 can potentially prevent PD-1 from shutting down the immune system, thus allowing immune cells to recognize and destroy cancer cells.

Gemcitabine is currently used to treat advanced or metastasized (spread) pancreatic cancer. It is used in patients whose disease cannot be removed by surgery and who have already been treated with other chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma with metastasis
* Must be off their prior cytotoxic regimen a minimum of two weeks but no more than four weeks from initiating trial treatment.

Measurable disease by RECIST 1.1.

Demonstrate adequate organ function

Normal Vitamin D level.

Able to submit an archival tumor specimen (primary or metastatic site). Patients with cytology only that do not have adequate archived tumor specimen available, will require a baseline biopsy.

Exclusion Criteria:

* Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 3 weeks of the first dose of trial treatment.
* Hypersensitivity to cabiralizumab, nivolumab, or gemcitabine or any of its excipients.
* Previous malignancies (except non-melanoma skin cancers, and in situ bladder, gastric, colorectal, endometrial, cervical/dysplasia, melanoma, or breast cancers) unless complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period.
* Evidence of central nervous system (CNS) metastasis
* Participants with active, known, or suspected autoimmune disease.
* Current or history of clinically significant muscle disorders (e.g., myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels.
* Uncontrolled or significant cardiovascular disease
* Prior organ allograft or allogeneic bone marrow transplantation.
* Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis.
* Evidence of coagulopathy or bleeding diathesis.
* Has received prior therapy with a CSF-1R pathway inhibitors, anti-PD-1, anti-PD-L1, anti PD-L2, anti-CTLA-4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hitendra Patel, MD, Principal Investigator — University of California, San Diego; Andrew Lowy, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine +Nivolumab + Cabiralizumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine +Nivolumab + Cabiralizumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Number of Participants Negative for PDL-1 [Count of Participants; unit: Participants] — Measurement of PDL-1: negative
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: To estimate Progression Free Survival (PFS rates) at 6 months per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Gemcitabine +Nivolumab + Cabiralizumab
Number analyzed (Participants) | 2
participants | 1

2. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Overall Survival (OS)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Gemcitabine +Nivolumab + Cabiralizumab
Number analyzed (Participants) | 2
participants | 1

ADVERSE EVENTS:
Time Frame: Through study completion (3 years & 8 months; 44 months)
Arm/Group | Gemcitabine +Nivolumab + Cabiralizumab
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine +Nivolumab + Cabiralizumab (N=2)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine +Nivolumab + Cabiralizumab (N=2)
Syncope (General disorders) | 1 (1)
Right flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated Creatinine Kinase (Metabolism and nutrition disorders) | 1 (2)
Thrombocytopenia - Grade 3 (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03697564/Prot_SAP_000.pdf